CLINICAL TRIAL: NCT02513576
Title: A Randomized, Controlled Study of Physiotherapy Exercises in Patients With Sternal Instability Due to Mediastinitis After Cardiovascular Surgery
Brief Title: Physiotherapy Exercises in Patients With Sternal Instability After Cardiovascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emilia Nozawa, PT PhD (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor-Investigator, Emilia Nozawa, PT PhD, principal investigator, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 51770
Record Dates: First submitted 2015-06-30; First posted 2015-07-31 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Mediastinitis; Coronary Artery Disease; Cardiovascular Infections
Keywords: Sternal instability; physical therapy; Respiratory muscle strength
MeSH Terms: conditions — Mediastinitis; Coronary Artery Disease; Cardiovascular Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physiotherapy exercises (Experimental): Two strategies of abdominal exercises with and without movement of the upper limbs applied in patients with sternal instability as randomization.
  Interventions: Other: physiotherapy exercises

INTERVENTIONS:
Other: physiotherapy exercises — Consisted of trunk stabilization exercises.The exercises were undertaken for 15 minutes every day for tree weeks. Patients were the contract their abdominal muscles with an emphasis on the transverse abdominal. Patients were to contract their abdominal muscles in a supine,sitting and stand up position.

SUMMARY:
Sternal instability caused by mediastinitis is one of the most feared complications for cardiac surgery team for generating large commitments and functional damages to patients. Biomechanically, the contraction of abdominal muscles such as transverse abdominal, produces forces that result in a "corset-like" action and anterior thoracic cage muscles too may assist in stabilizing the sternum. Thus, strengthening the abdominal muscles might contribute to the recovery of functional aspects. The aim was to evaluate whether contraction and strengthening the abdominal muscles could improve lung function and respiratory muscle strength in patients with sternal instability.

DETAILED DESCRIPTION:
Sternal instability was confirmed by physical examination and confirmed by chest tomography. The data were collected before and after the 3-week period of intervention.

Sternal instability way assessed by the unstable sternal scale, graduated from zero to 4 points.

The respiratory muscle strength was measured through Manuvacuometry and the pulmonary function by the spirometry.

Pain was recorded by using a Visual Analog Scale (0 -10); Discomfort Scale( 0-10) and Identification of Activities that cause pain and discomfort.

Patients underwent abdominal exercise protocol for three weeks once a day, lasting about 15 minutes followed by the physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative period of cardiovascular surgery by median sternotomy with sternal instability
* Written Inform consent

Exclusion Criteria:

* Chest Tube
* Hemodynamic instability
* Neurological alteration
* Active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Improvement of pulmonary function | 3 weeks
  Measure of maximal muscles respiratory pressures and spirometry tests

SECONDARY OUTCOMES:
Measure of pain on the Visual Analog Scale | 3 weeks
  Pain Visual Analog Scale
Discomfort - using Discomfort Scale | 3 weeks
  Activities using Discomfort Scale

CONTACTS AND LOCATIONS:
Overall Officials: EMILIA NOZAWA, PHD, Principal Investigator — University of Sao Paulo; Patricia O Almeida, PT, Study Chair — HEART INSTITUTE (INCOR) HOSPITAL DAS CLINICAS; Ludhmila A Hajjar, PHD, Study Chair — University of Sao Paulo; Filomena G Gallas, PHD, Study Chair — University of Sao Paulo; Cristiane D Goncalves, FT, Study Chair — HEART INSTITUTE (INCOR) HOSPITAL DAS CLINICAS; Maria Ignez Z Feltrim, PHD, Study Director — University of Sao Paulo

REFERENCES:
- [Result] El-Ansary D, Waddington G, Adams R. Control of separation in sternal instability by supportive devices: a comparison of an adjustable fastening brace, compression garment, and sports tape. Arch Phys Med Rehabil. 2008 Sep;89(9):1775-81. doi: 10.1016/j.apmr.2008.01.025. PMID 18760163
- [Result] El-Ansary D, Waddington G, Adams R. Relationship between pain and upper limb movement in patients with chronic sternal instability following cardiac surgery. Physiother Theory Pract. 2007 Sep-Oct;23(5):273-80. doi: 10.1080/09593980701209402. PMID 17934967
- [Result] El-Ansary D, Waddington G, Adams R. Trunk stabilisation exercises reduce sternal separation in chronic sternal instability after cardiac surgery: a randomised cross-over trial. Aust J Physiother. 2007;53(4):255-60. doi: 10.1016/s0004-9514(07)70006-5. PMID 18047460
- [Result] Gorlitzer M, Folkmann S, Meinhart J, Poslussny P, Thalmann M, Weiss G, Bijak M, Grabenwoeger M. A newly designed thorax support vest prevents sternum instability after median sternotomy. Eur J Cardiothorac Surg. 2009 Aug;36(2):335-9; discussion 339. doi: 10.1016/j.ejcts.2009.01.038. Epub 2009 Mar 9. PMID 19272785
- [Result] Fawzy H, Osei-Tutu K, Errett L, Latter D, Bonneau D, Musgrave M, Mahoney J. Sternal plate fixation for sternal wound reconstruction: initial experience (retrospective study). J Cardiothorac Surg. 2011 Apr 29;6:63. doi: 10.1186/1749-8090-6-63. PMID 21529357
- [Result] Lepelletier D, Poupelin L, Corvec S, Bourigault C, Bizouarn P, Blanloeil Y, Reynaud A, Duveau D, Despins P. Risk factors for mortality in patients with mediastinitis after cardiac surgery. Arch Cardiovasc Dis. 2009 Feb;102(2):119-25. doi: 10.1016/j.acvd.2008.11.003. Epub 2009 Feb 3. PMID 19303579
- [Result] Cowan KN, Teague L, Sue SC, Mahoney JL. Vacuum-assisted wound closure of deep sternal infections in high-risk patients after cardiac surgery. Ann Thorac Surg. 2005 Dec;80(6):2205-12. doi: 10.1016/j.athoracsur.2005.04.005. PMID 16305872
- [Result] Costa D, Goncalves HA, Lima LP, Ike D, Cancelliero KM, Montebelo MI. New reference values for maximal respiratory pressures in the Brazilian population. J Bras Pneumol. 2010 May-Jun;36(3):306-12. doi: 10.1590/s1806-37132010000300007. English, Portuguese. PMID 20625667
- [Result] Sakamoto H, Fukuda I, Oosaka M, Nakata H. Risk factors and treatment of deep sternal wound infection after cardiac operation. Ann Thorac Cardiovasc Surg. 2003 Aug;9(4):226-32. PMID 13129420
- [Result] Gelape CL. Surgical wound infection following heart surgery. Arq Bras Cardiol. 2007 Jul;89(1):e3-9. doi: 10.1590/s0066-782x2007001300013. No abstract available. English, Portuguese. PMID 17768574
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882